CLINICAL TRIAL: NCT04089397
Title: Randomized Open-label Trial Evaluating Light Therapy on Sleep Quality in Dialysis Patients
Brief Title: Light Therapy on Sleep Quality in Dialysis Patients
Acronym: LUMIDIAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Annecy Genevois (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-11-LUMIDIAL; 2018-A02276-49 (Other: ID-RCB)
Record Dates: First submitted 2019-09-11; First posted 2019-09-13 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2019-11

CONDITIONS: Chronic Renal Failure; Sleep Disorder; Hemodialysis; Light Therapy
Keywords: light therapy in sleep disorders of dialysis patients
MeSH Terms: conditions — Kidney Failure, Chronic; Sleep Wake Disorders | interventions — Phototherapy

STUDY DESIGN:
Intervention Model Description: Randomized open-label trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Light therapy group (Experimental): Five weeks of light therapy, with 3 weekly sessions of 30 minutes, to be performed between 8:00 to 10:00, the days of dialysis (at home, for patients dialyzing the afternoon, or during dialysis for patients dialyzing in the morning)
  Interventions: Device: Light Therapy
- Control group (No Intervention): Usual care, without light therapy

INTERVENTIONS:
Device: Light Therapy — Five weeks of light therapy, with 3 weekly sessions of 30 minutes, to be performed between 8:00 to 10:00, the days of dialysis
  Other Names: Lumie Brazil® (light therapy device for the treatment of seasonal affective disorders)
  Arms: Light therapy group

SUMMARY:
Sleep disorders are common in dialysis patients. At present, the management of insomnia in patients with chronic renal failure is not significantly different from that of the general population, which focuses on the management of co-factors, sleep hygiene, and cognitive-behavioral therapy.

Light therapy is a paramedical practice that involves exposing a patient to a light intensity greater than 5000 Lux (usually 10,000 Lux) for 30 minutes in the morning between 7:00 and 8:30. Its impact is partly mediated by an improvement in the nycthemeral cycle of melatonin.

Light therapy may improve sleep disorders and anxious-depressive elements as suggested in the literature. This technique has not yet been evaluated in dialysis patients, whereas easy to set up.

DETAILED DESCRIPTION:
Sleep disorders are common in dialysis patients. Indeed, several studies have reported that the prevalence of these disorders is higher than that of the general population. At present, the management of insomnia in patients with chronic renal failure is not significantly different from that of the general population, which focuses on the management of co-factors, sleep hygiene, and cognitive-behavioral therapy.

Light therapy is a paramedical practice that involves exposing a patient to a light intensity greater than 5000 Lux (usually 10,000 Lux) for 30 minutes in the morning between 7:00 and 8:30. Its impact is partly mediated by an improvement in the nycthemeral cycle of melatonin. Light therapy has been studied in several pathologies. In the context of renal insufficiency, only one randomized study was conducted in renal transplant patients: out of 30 patients, the effect of light therapy regained an 11-minute increase in sleep latency, an earlier awakening of 24 minutes, and a gain in the DASS-21 depression score of 1.7 points while there was no improvement in his three parameters in the control group. Interest in light therapy has also been evaluated in seasonal and non-seasonal depression. In a meta-analysis of 458 patients, light therapy adjuvant use was as effective as the addition of a second molecule.

Light therapy may improve sleep disorders and anxious-depressive elements as suggested in the literature. This technique has not yet been evaluated in dialysis patients, whereas easy to set up.

We therefore wish to set up a clinical study to determine whether a light therapy technique in the morning during dialysis or at home improves the quality of sleep of chronic hemodialysis patients. The secondary objectives will be to specify the improved sleep parameters, to evaluate the impact on the anxious-depressive score, the arterial hypertension, and the nutritional state, and the residual effect of light therapy.

The aim of this trial is to determine whether a light therapy technique in the morning during dialysis or at home improves the quality of sleep of chronic hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient in conventional hemodialysis or hemodiafiltration for at least 3 months
* Patient requiring a dialysis session three times a week in the investigational site
* Patient benefiting from a social security scheme
* Patient informed and having given his free and informed consent to participate in the study

Exclusion Criteria:

* Patient with binocular blindness and / or age-related macular degeneration
* Eye fatigue
* Patient who has undergone a recent eye surgery (less than 3 months) or for whom such an operation is planned in the next 20 weeks
* Patient taking medications known to be responsible for photosensitivity
* Pregnant or lactating woman
* Patient under guardianship or curatorship
* Patient unable to give free and informed consent

Exclusion during the study - premature stop

* Wishes of the patient or the physician
* Appearance of unexplained visual disturbances
* Kidney transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-05-11 (Actual); Study Completion 2020-05-11 (Actual)

PRIMARY OUTCOMES:
Impact of light therapy on the quality of sleep of dialysis patients | 5 weeks
  The Pittsburgh Sleep Quality Index (PSQI) questionnaire is a self-rated questionnaire designed to measure sleep quality and disturbance over the past month in clinical populations. The sleep component scores are summed to yield a total score ranging from 0 to 21 with the higher total score (referred to as global score) indicating worse sleep quality.
  The primary endpoint is the measured difference in PSQI score between baseline and 5 weeks post-exposure to light therapy between the two arms of the study (no light therapy versus active light therapy).

SECONDARY OUTCOMES:
Pathological sleep disorders defined by PSQI score > 5 | 5 weeks
  Percentage of patients with a PSQI score > 5 measured in both arms at baseline and after 5 weeks
Analysis of each component of the PSQI score | 5 weeks
  There are 7 components in the PSQI score (sleep duration, sleep disturbance, sleep latency, daytime dysfunction due to sleepiness, sleep efficiency, overall sleep quality, and sleep medication use). Each of the sleep components yields a score ranging from 0 to 3, with 3 indicating the greatest dysfunction.
  Difference of the medians obtained on each component of the PSQI score in both arms at baseline and after 5 weeks
Anxious-depressive state of the patients | 5 weeks
  The French Depression Anxiety Stress Scales (DASS 21) is a 21-item self-rated questionnaire designed to measure the emotional states of depression, anxiety and stress over the past week. The scale to which each item belongs is indicated by the letter D (Depression), A (Anxiety) and S (Stress). For each scale, scores are summed with the higher scores corresponding to the most severe status.
  Total score difference obtained from the questionnaire French Depression Anxiety Stress Scales (DASS 21) in both arms at baseline and after 5 weeks
Impact of light therapy on nutritional intake of patients | 10 weeks
  The normalized protein catabolic rate is a formula commonly used to assess dietary protein intake in dialysis patients, as a means towards determining nutritional adequacy.
  Absolute difference in Normalized Protein Catabolic Rate value in both arms at baseline, after 5 weeks and 10 weeks
Systolic Blood Pressure values | 10 weeks
  Absolute difference in systolic blood pressure in both arms at baseline, after 5 weeks and 10 weeks
Diastolic Blood Pressure values | 10 weeks
  Absolute difference in diastolic blood pressure in both arms at baseline, after 5 weeks and 10 weeks
Side effects of light therapy | 5 weeks
  Number and frequency of side effects
Impact of home care on the effectiveness of the primary endpoint | 5 weeks
  The Pittsburgh Sleep Quality Index (PSQI) questionnaire is a self-rated questionnaire designed to measure sleep quality and disturbance over the past month in clinical populations. The sleep component scores are summed to yield a total score ranging from 0 to 21 with the higher total score (referred to as global score) indicating worse sleep quality.
  Difference in the average PSQI score between the two subgroups: home care versus during dialysis light therapy
Evaluation of the residual duration of the effect of light therapy on sleep disorder | 5 weeks
  The Pittsburgh Sleep Quality Index (PSQI) questionnaire is a self-rated questionnaire designed to measure sleep quality and disturbance over the past month in clinical populations. The sleep component scores are summed to yield a total score ranging from 0 to 21 with the higher total score (referred to as global score) indicating worse sleep quality.
  Average difference in PSQI score at the end of the procedure and 5 weeks later.
Evaluation of the residual duration of the effect of light therapy on anxious-depressive state of the patients | 5 weeks
  The French Depression Anxiety Stress Scales (DASS 21) is a 21-item self-rated questionnaire designed to measure the emotional states of depression, anxiety and stress over the past week. The scale to which each item belongs is indicated by the letter D (Depression), A (Anxiety) and S (Stress). For each scale, scores are summed with the higher scores corresponding to the most severe status.
  Average difference in DASS 21 score, at the end of the procedure and 5 weeks later.

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Franko, MD, Principal Investigator — CH Annecy Genevois
Locations (1):
- CH Annecy Genevois, Pringy, France